CLINICAL TRIAL: NCT01451580
Title: A Phase II Study of Pegylated Liposomal Doxorubicin (Lipo-Dox) Combined With Cyclophosphamide /5-Fluorouracil as Second Line Chemotherapy in the Treatment of Metastatic Breast Cancer
Brief Title: Lipo-dox and Cyclophosphamide /5-Fluorouracil in Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TTY Biopharm (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: LD0411
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Phase II; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: Lipo-Dox

SUMMARY:
To determine the overall objective response rate of pegylated liposomal doxorubicin （Lipo-Dox）combined with cyclophosphamide/5-FU as second-line treatment in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proved breast cancer with metastatic disease

Exclusion Criteria:

* life expectancy less than 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Kun Chang, Principal Investigator — Chang Gung Memorial Hospital, Lin-Kou Medical Center
Locations (1):
- CGMH, Linko, Taiwan